CLINICAL TRIAL: NCT01659658
Title: A Phase 3, Randomized, Controlled, Open-label, Multicenter, Safety and Efficacy Study of Dexamethasone Plus MLN9708 or Physicians Choice of Treatment Administered to Patients With Relapsed or Refractory Systemic Light Chain (AL) Amyloidosis
Brief Title: Study of Dexamethasone Plus IXAZOMIB (MLN9708) or Physicians Choice of Treatment in Relapsed or Refractory Systemic Light Chain (AL) Amyloidosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C16011; 2011-005468-10 (EudraCT Number); U1111-1164-7621 (Registry Identifier: WHO); C16011-CTIL (Other: Israel); NL41603.028.12 (Registry Identifier: CCMO); 12/LO/1771 (Registry Identifier: NRES); MOH_2017-05-07_000374 (Other: CRS)
Record Dates: First submitted 2012-08-02; First posted 2012-08-08 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory Systemic Light Chain Amyloidosis
Keywords: MLN9708; Amyloidosis; Light Chain; IXAZOMIB; Tourmaline AL1; Drug Therapy
MeSH Terms: conditions — Recurrence; Amyloidosis | interventions — ixazomib; Dexamethasone; Melphalan; Cyclophosphamide; Thalidomide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Ixazomib + Dexamethasone (Experimental): Ixazomib 4 mg, capsules, orally, once on Days 1, 8, and 15 and dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle for up to a maximum of 95.2 months. Dexamethasone was increased up to 40 mg/day after 4 weeks, if tolerated.
  Interventions: Drug: IXAZOMIB; Drug: Dexamethasone
- Arm B: Dexamethasone + Melphalan (Active Comparator): Participants received dexamethasone 20 mg, orally, and melphalan 0.22 mg/kg, orally once on Days 1 through 4 of each 28-day cycle, for up to a maximum of 72.4 months.
  Interventions: Drug: Dexamethasone; Drug: Melphalan
- Arm B: Dexamethasone + Cyclophosphamide (Active Comparator): Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22, and cyclophosphamide 500 mg, orally, on Days 1, 8 and 15 of each 28-day cycle for up to a maximum of 72.4 months.
  Interventions: Drug: Dexamethasone; Drug: Cyclophosphamide
- Arm B: Dexamethasone + Thalidomide (Active Comparator): Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15 and 22 of each 28-day cycle, and thalidomide daily at a starting dose of 50 mg and increased, as tolerated, to a maximum of 200 mg, orally for up to a maximum of 72.4 months.
  Interventions: Drug: Dexamethasone; Drug: Thalidomide
- Arm B: Dexamethasone + Lenalidomide (Active Comparator): Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15 and 22 of each 28-day cycle and lenalidomide 15 mg, orally, once on Days 1 through 21 every 28 days for up to a maximum of 72.4 months.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide

INTERVENTIONS:
Drug: IXAZOMIB — IXAZOMIB capsules
  Other Names: MLN9708
  Arms: Arm A: Ixazomib + Dexamethasone
Drug: Dexamethasone — Dexamethasone tablets
Drug: Melphalan — Melphalan tablets
  Arms: Arm B: Dexamethasone + Melphalan
Drug: Cyclophosphamide — Cyclophosphamide tablets
  Arms: Arm B: Dexamethasone + Cyclophosphamide
Drug: Thalidomide — Thalidomide capsules
  Arms: Arm B: Dexamethasone + Thalidomide
Drug: Lenalidomide — Lenalidomide capsules
  Arms: Arm B: Dexamethasone + Lenalidomide

SUMMARY:
The purpose of this study is to provide continued access of ixazomib and/or other study medications and to continue collecting relevant safety data to monitor participant's safety, determine whether dexamethasone plus IXAZOMIB improves hematologic response, 2-year vital organ (that is, heart or kidney) deterioration and mortality rate versus a physician's choice of a chemotherapy regimen in participants diagnosed with relapsed or refractory systemic light chain (AL) amyloidosis.

DETAILED DESCRIPTION:
The drug being tested in this study is called IXAZOMIB. IXAZOMIB was being tested to treat people who have relapsed or Refractory Systemic Light Chain (AL) Amyloidosis.

The study will enroll approximately 177 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* IXAZOMIB 4 mg plus Dexamethasone 20 mg
* Physician's choice: Participants will receive one of the following treatment options as selected by the physician:

  1. Dexamethasone 20 mg
  2. Dexamethasone 20 mg + Melphalan 0.22 mg/kg
  3. Dexamethasone 20 mg + Cyclophosphamide 500 mg
  4. Dexamethasone 20 mg + Thalidomide 200 mg
  5. Dexamethasone 20 mg + Lenalidomide 15 mg
  6. All participants will be asked to take oral formulation of the drugs. In both treatment arms, each participant will continue to receive sequential cycles of therapy until disease progression, unacceptable toxicity, or until the study is terminated, whichever occurs first. Participants in Arm B receiving melphalan and dexamethasone will be treated to best response plus 2 additional cycles.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 120 months (10 years), including 84 months of enrollment and 36 months of follow-up after the last participant is enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years or older.
2. Biopsy-proven diagnosis of primary systemic light chain amyloidosis (AL amyloidosis) according to the following standard criteria:

   1. Histochemical diagnosis of amyloidosis, as based on tissue specimens with Congo red staining with exhibition of an apple-green birefringence
   2. If clinical and laboratory parameters insufficient to establish AL amyloidosis or in cases of doubt, amyloid typing may be necessary.
3. Measurable disease as defined by serum differential free light chain concentration (dFLC, difference between amyloid forming [involved] and nonamyloid forming [uninvolved] free light chain [FLC]) ≥ 50 mg/L.
4. Objective, measurable major (cardiac or renal) organ amyloid involvement as defined as follows (amyloid involvement of at least 1 required):

   1. Cardiac involvement is defined as the presence of a mean left ventricular wall thickness on echocardiogram greater than 12 mm in the absence of other potential causes of left ventricular hypertrophy (controlled hypertension is allowed) with a noncardiac biopsy showing amyloid, or a positive cardiac biopsy in the presence of clinical or laboratory evidence of involvement. If there is isolated cardiac involvement, then typing of amyloid deposits is recommended.
   2. Renal involvement is defined as proteinuria (predominantly albumin) >0.5 g/day in a 24-hour urine collection.

   Note: Amyloid involvement of other organ systems is allowed, but not required.
5. Must be relapsed or refractory after 1 or 2 prior therapies. For this protocol, relapsed is defined as progressive disease (PD) documented more than 60 days after last dose; refractory is defined as documented absence of hematologic response or hematologic progression on or within 60 days after last dose of prior therapy.

   1. Participant must not have been previously treated with proteasome inhibitors. (The sponsor reserves the right to open the study to proteasome inhibitor-exposed participants in the future, at some time point after the first interim analysis (IA). In that case, the participant may not be refractory to proteasome inhibitor therapy.)
   2. Given that the physician may select from an offered list of regimens to treat a specific participant, the participant may be refractory to an agent/s listed within the list of offered treatment choices
   3. Must have recovered (ie, ≤ Grade 1 toxicity or participant's baseline status) from the reversible effects of prior therapy
   4. If a participant has received a transplant as his/her first-line therapy, he/she must be at least 3 months post transplantation and recovered from the side effects of the stem cell transplant.
6. Must meet criteria for 1 of the following AL Amyloidosis Risk Stages (as defined by N-terminal proBNP [NT-proBNP] cut-off of < 332 pg/mL and troponin T cut-off of 0.035 ng/mL as thresholds):

   1. Stage 1: both NT-proBNP and troponin T under threshold
   2. Stage 2: either NT-proBNP or troponin T (but not both) over threshold;
   3. Stage 3: both NT-proBNP and troponin T over threshold (but NT-proBNP < 8000 pg/mL)
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
8. Clinical laboratory values:

   1. Absolute neutrophil count ≥ 1000/µL
   2. Platelet count ≥ 75,000/µL
   3. Total bilirubin ≤ 1.5 upper limit of normal (ULN), except for participants with Gilbert's syndrome as defined by > 80% unconjugated bilirubin and total bilirubin ≤ 6 mg/dL
   4. Alkaline phosphatase ≤ 5 x ULN
   5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 x ULN
   6. Calculated creatinine clearance ≥ 30 mL/min
9. Female participants who:

   1. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study treatment, AND
   2. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   3. Agree to practice true abstinence when this is line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.).

   Male participants, even if surgically sterilized (ie, status post vasectomy), who:
   1. Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, AND
   2. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   3. Agree to practice true abstinence when this is line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
10. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

1. Amyloidosis due to mutations of the transthyretin gene or presence of other non-AL amyloidosis.
2. Female participants who are lactating, breast feeding, or pregnant.
3. Medically documented cardiac syncope, uncompensated New York Heart Association (NYHA) Class 3 or 4 congestive heart failure, myocardial infarction within the previous 6 months, unstable angina pectoris, clinically significant repetitive ventricular arrhythmias despite antiarrhythmic treatment, or severe orthostatic hypotension or clinically important autonomic disease.
4. Clinically overt multiple myeloma, according to the International Myeloma Working Group (IMWG) criteria with at least 1 of the following:

   1. Bone lesions
   2. Hypercalcemia, defined as a calcium of > 11 mg/dL
5. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
6. Requirement for other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered to be investigational or which would be considered as a treatment of AL amyloidosis. However, participants may be on chronic steroids (maximum dose 20 mg/day prednisone or equivalent) if they are being given for disorders other than amyloidosis (eg, adrenal insufficiency, rheumatoid arthritis, etc.).
7. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
8. Ongoing or active infection, known human immunodeficiency virus (HIV) positive, active hepatitis B or C infection.
9. Psychiatric illness/social situations that would limit compliance with study requirements.
10. Known allergy to boron, MLN9708, any of the study treatments, their analogues, or excipients.
11. Systemic treatment with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment.
12. Diagnosed or treated for another malignancy within 3 years (or 5 years for participants in France) before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2012-12-26 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (66):
- United States (15):
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Brazil (5):
  - Centro de Pesquisas Oncologicas, Florianópolis, Santa Catarina
  - Hospital Universitario Clementino Fraga Filho (UFRJ), Rio de Janeiro
  - Irmandade Da Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Ostrava, Ostrava, Moravskoslezsk Kraj
  - Vseobecna fakultni nemocnice v Praze, Prague, Praha, Hlavni Mesto
- Denmark (2):
  - Arhus Universitetshospital Arhus Sygehus, Aahus
  - Rigshospitalet, Copenhagen
- France (5):
  - Hotel Dieu, Nantes, Loire-Atlantique
  - Hopital Claude Huriez, Lille
  - Centre Hospitalier et Universitaire de Limoges, Limoges
  - Hopital Saint Louis, Paris
  - Hopital de Rangueil, Toulouse
- Germany (3):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Hamburg Eppendorf, Hamburg
  - Universitat Heidelberg, Heidelberg
- Greece (2):
  - University General Hospital of Patras, Pátrai, Achaia
  - Alexandra Hospital, Athens
- Israel (5):
  - Rambam Health Corporation, Haifa
  - Hadasit Medical Research Services and Development Ltd, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - PPDS, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (2):
  - Institute of Hematology "Seragnoli" University of Bologna, Bologna
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam, North Holland
  - Maastricht University Medical Center, AZ Maastricht
  - Universitair Medisch Centrum Utrecht, Utrecht
- South Korea (5):
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital at Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St Mary's Hospital, Seoul
- Spain (5):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Free and University College Medical School, London
  - Manchester Royal Infirmary, Manchester
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Sanchorawala V, Wechalekar AD, Kim K, Schonland SO, Landau HJ, Kwok F, Suzuki K, Dispenzieri A, Merlini G, Comenzo RL, Cherepanov D, Hayden VC, Kumar A, Labotka R, Faller DV, Kastritis E. Quality of life and symptoms among patients with relapsed/refractory AL amyloidosis treated with ixazomib-dexamethasone versus physician's choice. Am J Hematol. 2023 May;98(5):720-729. doi: 10.1002/ajh.26866. Epub 2023 Feb 14. PMID 36708469
- [Derived] Sanchorawala V, Palladini G, Kukreti V, Zonder JA, Cohen AD, Seldin DC, Dispenzieri A, Jaccard A, Schonland SO, Berg D, Yang H, Gupta N, Hui AM, Comenzo RL, Merlini G. A phase 1/2 study of the oral proteasome inhibitor ixazomib in relapsed or refractory AL amyloidosis. Blood. 2017 Aug 3;130(5):597-605. doi: 10.1182/blood-2017-03-771220. Epub 2017 May 26. PMID 28550039
- See also: To obtain more information on the study, click this link. — https://www.clinicaltrials.takeda.com/study-detail/5f6b601f4db2bf003ab49533??page=1&idFilter=C16011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 66 investigative sites from 12 December 2012 to 11 July 2022. The study was prematurely terminated based on the Sponsor's decision following the first interim analysis.
Pre-assignment Details: Participants with a diagnosis of relapsed or refractory (R/R) systemic light chain amyloidosis (AL) were enrolled in the study to receive ixazomib capsules or physician's choice of therapy, which included dexamethasone tablets alone or in combination with either melphalan, cyclophosphamide, thalidomide or lenalidomide.
Groups:
- Arm A: Ixazomib + Dexamethasone: Participants received ixazomib 4 mg, capsules, orally, once on Days 1, 8, and 15 and dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle for up to a maximum of 95.2 months. Dexamethasone was increased up to 40 mg/day after 4 weeks, if tolerated.
- Arm B: Dexamethasone + Cyclophosphamide: Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22, and cyclophosphamide 500 mg, orally, on Days 1, 8, and 15 of each 28-day cycle for up to a maximum of 72.4 months.
- Arm B: Dexamethasone + Thalidomide: Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle, and thalidomide daily at a starting dose of 50 mg and increased, as tolerated, to a maximum of 200 mg, orally for up to a maximum of 72.4 months.
- Arm B: Dexamethasone + Lenalidomide: Participants received dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle and lenalidomide 15 mg, orally, once on Days 1 through 21 every 28 days for up to a maximum of 72.4 months.
Period: Overall Study
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan | Arm B: Dexamethasone + Cyclophosphamide | Arm B: Dexamethasone + Thalidomide | Arm B: Dexamethasone + Lenalidomide
Started | 90 | 26 | 10 | 2 | 49
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 90 | 26 | 10 | 2 | 49
Not completed — Withdrawal by Patient | 18 | 4 | 2 | 0 | 11
Not completed — Study Terminated by Sponsor | 9 | 7 | 0 | 1 | 4
Not completed — Reason not Specified | 61 | 15 | 8 | 1 | 34
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan | Arm B: Dexamethasone + Cyclophosphamide | Arm B: Dexamethasone + Thalidomide | Arm B: Dexamethasone + Lenalidomide | Total
Number analyzed (Participants) | 90 | 26 | 10 | 2 | 49 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.83) | 64.8 (8.73) | 60.0 (14.97) | 65.0 (2.83) | 64.9 (8.68) | 63.9 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 11 | 4 | 2 | 22 | 74
  Male | 55 | 15 | 6 | 0 | 27 | 103
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 2 | 3
  Not Hispanic or Latino | 85 | 25 | 9 | 2 | 40 | 161
  Unknown or Not Reported | 5 | 0 | 1 | 0 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 16 | 9 | 5 | 1 | 1 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1
  White | 70 | 17 | 5 | 1 | 48 | 141
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 5 | 0 | 1 | 0 | 3 | 9
  United States | 24 | 2 | 3 | 0 | 13 | 42
  Czechia | 2 | 0 | 0 | 0 | 1 | 3
  Denmark | 0 | 0 | 0 | 1 | 2 | 3
  France | 3 | 1 | 0 | 0 | 1 | 5
  Germany | 8 | 5 | 0 | 0 | 3 | 16
  United Kingdom | 10 | 4 | 0 | 0 | 3 | 17
  Greece | 6 | 0 | 2 | 0 | 7 | 15
  Italy | 3 | 0 | 0 | 0 | 4 | 7
  Netherlands | 3 | 1 | 0 | 0 | 0 | 4
  Spain | 1 | 1 | 0 | 0 | 3 | 5
  Turkey | 1 | 0 | 0 | 0 | 0 | 1
  Australia | 8 | 0 | 0 | 0 | 6 | 14
  Brazil | 0 | 0 | 0 | 1 | 0 | 1
  China | 4 | 2 | 0 | 0 | 0 | 6
  Israel | 3 | 3 | 0 | 0 | 2 | 8
  Japan | 2 | 5 | 0 | 0 | 0 | 7
  Korea, Republic of | 7 | 2 | 4 | 0 | 1 | 14
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed is the number of participants with data available for height.
  centimeters (cm)
    number analyzed (Participants) | 90 | 26 | 10 | 2 | 48 | 176
    (all) | 170.40 (10.507) | 167.07 (8.662) | 170.65 (13.274) | 160.50 (13.435) | 169.17 (10.532) | 169.48 (10.444)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 77.33 (16.740) | 70.95 (12.476) | 70.20 (21.815) | 50.10 (15.415) | 75.35 (17.144) | 75.13 (16.830)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Hematologic Response
Description: Overall hematologic response was defined as the percentage of participants with complete response (CR), very good partial response (VGPR) and partial response (PR) based on central laboratory results and the 2010 International Society of Amyloidosis (ISA) Consensus Criteria as assessed by an adjudication committee. CR: Complete disappearance of M-protein from serum and urine on immunofixation, and normalization of free light chain (FLC) ratio. VGPR: differential free light chain (difference between involved and uninvolved FLC levels; dFLC) < 40 mg/L. PR: ≥50% reduction in dFLC. Percentages were rounded off to the nearest decimal.
Time Frame: From first dose of study drug until discontinuation of study drug due to disease progression or unacceptable toxicity, or death whichever occurs first (up to 115 months)
Population: ITT Population included all participants who were randomized. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan | Arm B: Dexamethasone + Cyclophosphamide | Arm B: Dexamethasone + Thalidomide | Arm B: Dexamethasone + Lenalidomide
Number analyzed (Participants) | 85 | 24 | 10 | 2 | 47
percentage of participants | 53 [41.8 to 63.9] | 58 [36.6 to 77.9] | 30 [6.7 to 65.2] | 50 [1.3 to 98.7] | 51 [36.1 to 65.9]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan vs Arm B: Dexamethasone + Cyclophosphamide vs Arm B: Dexamethasone + Thalidomide vs Arm B: Dexamethasone + Lenalidomide; Statistical analysis was planned to be collected and analyzed in a combined manner for the non-ixazomib arm groups versus ixazomib group in this outcome measure; Test type: Superiority; p = 0.7623, Cochran-Mantel-Haenszel — P-value was calculated from the unstratified Cochran-Mantel-Haenszel (CMH) test to compare hematologic response rate between the treatment arms; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.60 to 2.01] — Odds ratio was derived from a logistic regression model with treatment and 95% confidence interval (CI) for the odds ratio was based on the Wald approximation

2. Primary Outcome: 2-Year Vital Organ (Heart or Kidney) Deterioration and Mortality Rate
Description: Cardiac (Heart) deterioration was defined as the need for hospitalization for heart failure. Kidney deterioration was defined as progression to end-stage renal disease (ESRD) with the need for maintenance dialysis or renal transplantation. Vital organ deterioration was evaluated by an adjudication committee. Percentages were rounded off to the nearest decimal. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: Up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide: Participants received dexamethasone 20 mg, orally, and melphalan 0.22 mg/kg, orally once on Days 1 through 4 of each 28-day cycle, for up to a maximum of 72.4 months OR dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22, and cyclophosphamide 500 mg, orally, on Days 1, 8, and 15 of each 28-day cycle for up to a maximum of 72.4 months OR dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle, and thalidomide daily at a starting dose of 50 mg and increased, as tolerated, to a maximum of 200 mg, orally for up to a maximum of 72.4 months OR dexamethasone 20 mg, orally, once weekly on Days 1, 8, 15, and 22 of each 28-day cycle and lenalidomide 15 mg, orally, once on Days 1 through 21 every 28 days for up to a maximum of 72.4 months.
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 85 | 83
percentage of participants | 47 [36.1 to 58.2] | 54 [41.7 to 64.1]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.3510, Cochran-Mantel-Haenszel — P-value was calculated from the unstratified CMH test to make comparisons between the 2 treatment arms; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.41 to 1.38] — Odds ratio was derived from a logistic regression model with treatment and 95% CI for the odds ratio was based on the Wald approximation

3. Secondary Outcome: Percentage of Participants With Complete Hematologic Response
Description: Complete hematologic response was defined as the percentage of participants with CR based on central laboratory results and the 2010 ISA Consensus Criteria as assessed by the investigator. CR: Complete disappearance of M-protein from serum and urine on immunofixation, and normalization of FLC ratio. Percentages were rounded off to the nearest decimal. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
percentage of participants | 30 [20.8 to 40.6] | 17 [10.0 to 26.8]

4. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 69.55 [0.8 to 95.5] | 43.17 [0.0 to 82.4]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.389, Log Rank — P-value was calculated using log-rank test stratified by the stratification factors; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.52 to 1.29]; Unadjusted stratified Cox regression model was used to estimate the hazard ratio and its 95% CIs for the treatment effect using the stratification factors

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of first documentation of hematologic disease progression, or organ (cardiac or renal) progression, or death due to any cause, whichever occurred first according to central laboratory results and ISA criteria as evaluated by the investigator. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 11.86 [0.8 to 72.0] | 7.62 [0.0 to 71.1]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.135, Log Rank — P-value was calculated using stratified log-rank test with stratification factors; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.52 to 1.09]; [other analysis details as in outcome 4, analysis 1]

6. Secondary Outcome: Hematologic Disease Progression Free Survival
Description: Hematologic disease PFS was defined as the time from the date of randomization to the date of first documentation of hematologic PD according to central laboratory results and ISA criteria as evaluated by an adjudication committee, or death due to any cause, whichever occurred first. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 85 | 83
months | 29.50 [0.1 to 54.5] | 27.73 [0.1 to 43.5]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.2421, Log Rank — P-value was calculated using log-rank test stratified by the stratification factors; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.48 to 1.21]; [other analysis details as in outcome 4, analysis 1]

7. Secondary Outcome: Time to Vital Organ (Heart or Kidney) Deterioration and Mortality Rate
Description: Time to vital organ deterioration or death was assessed by the investigator and defined as the time from randomization to vital organ (heart or kidney) deterioration or death, whichever occurs first. Cardiac deterioration is defined as the need for hospitalization for heart failure. Kidney deterioration is defined as progression to ESRD with the need for maintenance dialysis or renal transplantation. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: From randomization to time of vital organ deterioration or death (up to 115 months)
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 38.67 [0.0 to 70.5] | 26.09 [0.0 to 71.1]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.036, Log Rank — P-value was calculated using log-rank test stratified by the stratification factors; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.39 to 0.97]; [other analysis details as in outcome 4, analysis 1]

8. Secondary Outcome: Percentage of Participants With Best Vital Organ (Cardiac and/or Kidney) Response
Description: Vital organ (heart and kidney) response rate was defined as the percentage of participants who achieved vital organ response according to central laboratory results and ISA criteria as evaluated by an adjudication committee. A vital organ response was defined as response of 1 or 2 of the involved vital organs with no change from Baseline in the rest of involved vital organs. Percentages were rounded off to the nearest decimal. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 85 | 83
percentage of participants | 19 [11.2 to 28.8] | 12 [5.9 to 21.0]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.2260, Cochran-Mantel-Haenszel — P-value was calculated from the unstratified CMH test to compare vital organ response rate between the 2 treatment arms; Odds Ratio (OR) = 1.69, 95% CI 2-sided [0.72 to 3.99] — Odds ratio was calculated from a logistic regression model with treatment and 95% CI for the odds ratio was based on the Wald approximation

9. Secondary Outcome: Vital Organ Progression Free Survival
Description: Vital organ PFS is defined as the time from the date of randomization to the date of first documentation of progression of vital organ (heart or kidney) according to central laboratory results and ISA criteria as evaluated by an adjudication committee, or death due to any cause, whichever occurs first. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 15.77 [0.0 to 72.0] | 11.01 [0.0 to 71.1]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.163, Log Rank — P-value was calculated using stratified log-rank test with stratification factors; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.52 to 1.12] — Unadjusted stratified Cox regression model was used to estimate the hazard ratio and its 95% CIs for the treatment effect using the stratification factors

10. Secondary Outcome: Duration of Hematologic Response
Description: Duration of hematologic response (DOR) was defined as the time from the date of first documentation of a hematologic response to the date of first documented hematologic disease progression as determined by the investigator. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: From time of first documented response to disease progression (up to 115 months)
Population: ITT Population included all participants who were randomized. Overall number of participants analyzed is the number of hematologic responders.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 49 | 45
months | NA [1.8 to 71.1] — Median was not estimable due to excess amount of censoring among the participants for the analysis. | 21.19 [0.0 to 69.0]

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of an existing hospitalization, resulted in persistent or significant disability or incapacity, was a congenital anomaly/birth defect or medically important event.
Time Frame: From first dose of study drug through 30 days after administration of the last dose of study drug (up to 115 months)
Population: Safety Population included all participants who received at least 1 dose of any treatment drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan | Arm B: Dexamethasone + Cyclophosphamide | Arm B: Dexamethasone + Thalidomide | Arm B: Dexamethasone + Lenalidomide
Number analyzed (Participants) | 90 | 26 | 10 | 1 | 47
Participants | 44 | 11 | 2 | 0 | 17

12. Secondary Outcome: Time To Treatment Failure (TTF)
Description: TTF was defined as the time from randomization to the date of first documented treatment failure. Treatment failure was defined as: 1) death due to any cause; 2) hematologic progression or major organ progression according to central laboratory results and ISA criteria as evaluated by the investigator; 3) clinically morbid organ disease requiring additional therapy; or 4) withdrawn for any reason. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: ITT Population included all participants who were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 10.32 [7.52 to 14.82] | 5.32 [4.14 to 7.82]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.025, Log Rank — P-value was calculated using stratified log-rank test with stratification factors; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.49 to 0.96]; [other analysis details as in outcome 4, analysis 1]

13. Secondary Outcome: Time To Subsequent Anticancer Treatment
Description: Time to subsequent anticancer therapy was defined as the time from randomization to the first date of subsequent anticancer therapy. Participants without subsequent anticancer therapy were censored at the date of death or last known to be alive. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: From first dose of study drug until subsequent anticancer treatment (up to 115 months)
Population: ITT Population included all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 90 | 87
months | 26.48 [0.8 to 95.5] | 12.45 [0.0 to 72.7]
Statistical Analysis 1: Comparison: Arm A: Ixazomib + Dexamethasone vs Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide; Test type: Superiority; p = 0.010, Log Rank — P-value was calculated using stratified log-rank test with stratification factors; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.38 to 0.88]; [other analysis details as in outcome 4, analysis 1]

14. Secondary Outcome: Change From Baseline in 36-item Short Form General Health Survey (SF-36) Mental Component Summary Score at Week 28 of the PFS Follow-up
Description: SF-36 Version 2 is a multipurpose, participant completed, short-form health survey with 36 questions that consists of an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures. Physical component summary (PCS) is mostly contributed by physical function (PF), role physical (RP), bodily pain (BP), and general health (GH). Mental component summary (MCS) is mostly contributed by mental health (MH), role emotional (RE), social function (SF), and vitality (VT). Each component on the SF-36 item health survey is scored from 0 (best) to 100 (worst). Total score ranges from 0-100, where higher scores are associated with less disability and better quality of life. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: Baseline, Week 28 of the PFS Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
score on a scale |  | 2.0 (NA) — Standard deviation (SD) was not estimable for 1 participant.

15. Secondary Outcome: Change From Baseline in SF-36 Physical Component Summary Score at Week 28 of the PFS Follow-up
Description: as for outcome 14
Time Frame: Baseline, Week 28 of the PFS Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
score on a scale |  | 10.3 (NA) — SD was not estimable for 1 participant.

16. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-Ntx) Score at Week 28 of the PFS Follow-up
Description: The FACT/GOG-Ntx is a participant completed questionnaire that comprises 11 individual items evaluating symptoms of neurotoxicity on a 5-point scale where: 0=not at all (best) to 4=very much for a total possible score of 0 to 44. Symptom scores are inverted so that higher scores of FACT/GOG-Ntx indicate higher quality of life or functioning. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: Baseline, Week 28 of the PFS Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
score on a scale |  | 0.0 (NA) — SD was not estimable for 1 participant.

17. Secondary Outcome: Change From Baseline in Amyloidosis Symptom Scale Total Score at Week 28 of the PFS Follow-up
Description: The amyloidosis symptom scale questionnaire is a participant completed questionnaire that evaluates symptom severity of 3 symptoms: Swelling, Shortness of Breath and Dizziness, each rated on an 11-point scale where: 0=no symptoms to 10=very severe symptoms. Higher scores indicate worsening of symptoms. Total Score is the sum of all responses from the amyloidosis symptom scale ranging from 0 to 30. Higher scores represent higher levels of symptomatology or problems and a negative change from baseline indicates improvement. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: Baseline, Week 28 of the PFS Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
score on a scale |  | -16.0 (NA) — SD was not estimable for 1 participant.

18. Secondary Outcome: Number of Participants in Each Category of the EuroQol 5-Dimensional (EQ-5D) Questionnaire Score
Description: The European Quality of Life (EuroQOL) 5-Dimensional (EQ-5D) is a patient completed questionnaire consisting of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 3 possible choices: no problems to extreme problems. Higher scores=worsening of the quality of life. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: At Week 28 of the OS follow-up
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
Participants
  Mobility: No Problems in Walking About | 0 | 0
  Mobility: Some Problem in Walking About | 0 | 1
  Mobility: Confined to Bed | 0 | 0
  Self-Care: No Problems With Self- Care | 0 | 0
  Self-Care: Some Problems Washing or Dressing | 0 | 1
  Self-Care: Unable to Wash or Dress | 0 | 0
  Usual Activities: No Problems With Performing Usual Activities | 0 | 0
  Usual Activities: Some Problem With Performing Usual Activities | 0 | 1
  Usual Activities: Unable to Performing Usual Activities | 0 | 0
  Pain/Discomfort: No Pain or Discomfort | 0 | 0
  Pain/Discomfort: Moderate Pain or Discomfort | 0 | 1
  Pain/Discomfort: Extreme Pain or Discomfort | 0 | 0
  Anxiety/Depression: Not Anxious or Depressed | 0 | 0
  Anxiety/Depression: Moderately Anxious or Depressed | 0 | 0
  Anxiety/Depression: Extremely Anxious or Depressed | 0 | 1

19. Secondary Outcome: EuroQol 5-Dimension 3-Level (EQ-5D-3L) Visual Analogue Scale Score
Description: The EQ visual analogue scale (VAS) records the participant's self-rated health on a 20 centimeter vertical VAS that ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). Baseline is defined as the value collected at the time closest to, but prior to, the start of study drug administration. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: At Week 28 of the OS follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 0 | 1
score on a scale |  | 23.0 (NA) — SD was not estimable for 1 participant.

20. Secondary Outcome: Plasma Concentration of Ixazomib
Description: As prespecified in the protocol, data for this outcome measure was planned to be collected for ixazomib arm group only.
Time Frame: Cycle 1, Day 1: 1, 4 hours postdose, Day 14: 144 hours postdose; Cycle 2, Day 1: predose, Day 14: 144 hours postdose; Cycles 3 to 10, Day 1: predose (cycle length=28 days)
Population: Pharmacokinetic (PK) Analysis Population included participants with at least one PK sample that was collected and analyzed. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Arm A: Ixazomib + Dexamethasone
Number analyzed (Participants) | 78
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1: 1 Hour Post-dose: number analyzed (Participants) | 77
  Cycle 1 Day 1: 1 Hour Post-dose | 16.518 (97.0462)
  Cycle 1 Day 14: 4 Hours Post-dose | 10.652 (121.7231)
  Cycle 1 Day 14: 144 Hours Post-dose: number analyzed (Participants) | 73
  Cycle 1 Day 14: 144 Hours Post-dose | 3.875 (100.3055)
  Cycle 2 Day 1: Pre-dose: number analyzed (Participants) | 70
  Cycle 2 Day 1: Pre-dose | 2.000 (59.4061)
  Cycle 2 Day 14: 144 Hours Post-dose: number analyzed (Participants) | 60
  Cycle 2 Day 14: 144 Hours Post-dose | 4.726 (115.5653)
  Cycle 3 Day 1: Pre-dose: number analyzed (Participants) | 65
  Cycle 3 Day 1: Pre-dose | 2.187 (59.1378)
  Cycle 4 Day 1 Pre-dose: number analyzed (Participants) | 59
  Cycle 4 Day 1 Pre-dose | 2.276 (59.3690)
  Cycle 5 Day 1 Pre-dose: number analyzed (Participants) | 56
  Cycle 5 Day 1 Pre-dose | 2.264 (54.8881)
  Cycle 6 Day 1: Pre-dose: number analyzed (Participants) | 54
  Cycle 6 Day 1: Pre-dose | 2.235 (60.4723)
  Cycle 7 Day 1: Pre-dose: number analyzed (Participants) | 45
  Cycle 7 Day 1: Pre-dose | 2.299 (53.7147)
  Cycle 8 Day 1: Pre-dose: number analyzed (Participants) | 43
  Cycle 8 Day 1: Pre-dose | 2.038 (58.6811)
  Cycle 9 Day 1: Pre-dose: number analyzed (Participants) | 42
  Cycle 9 Day 1: Pre-dose | 2.143 (55.0715)
  Cycle 10 Day 1: Pre-dose: number analyzed (Participants) | 42
  Cycle 10 Day 1: Pre-dose | 2.232 (57.4067)

21. Secondary Outcome: Number of Hospitalizations
Description: A hospitalization was defined as at least one overnight stay in an intensive care unit and/or non-intensive care unit. If a single hospitalization included both an intensive care unit stay and a non-intensive care unit stay, the hospitalization was counted only once (as an intensive care unit stay). The mean number of hospitalizations is reported in this outcome measure. As prespecified in the protocol, data was planned to be collected and analyzed in a combined way for non-ixazomib arm groups in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan/Cyclophosphamide/Thalidomide/Lenalidomide
Number analyzed (Participants) | 85 | 83
hospitalizations | 1.8 (1.34) | 1.4 (0.80)

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after administration of the last dose of study drug (up to 115 months)
Description: All-cause mortality: ITT Population included all participants who were randomized. Serious and other adverse events: Safety Population included all participants who received at least 1 dose of any treatment drug.
Arm/Group | Arm A: Ixazomib + Dexamethasone | Arm B: Dexamethasone + Melphalan | Arm B: Dexamethasone + Cyclophosphamide | Arm B: Dexamethasone + Thalidomide | Arm B: Dexamethasone + Lenalidomide
All-Cause Mortality (participants affected / at risk) | 40/90 | 14/26 | 4/10 | 0/2 | 22/49
Serious Adverse Events (participants affected / at risk) | 44/90 | 11/26 | 2/10 | 0/1 | 17/47
Other Adverse Events (participants affected / at risk) | 86/90 | 24/26 | 9/10 | 1/1 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ixazomib + Dexamethasone (N=90) | Arm B: Dexamethasone + Melphalan (N=26) | Arm B: Dexamethasone + Cyclophosphamide (N=10) | Arm B: Dexamethasone + Thalidomide (N=1) | Arm B: Dexamethasone + Lenalidomide (N=47)
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cardiac amyloidosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 3 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Herpes zoster cutaneous disseminated (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Jaw cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 4 | 0 | 0 | 2
Pneumonia chlamydial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal cord infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Ixazomib + Dexamethasone (N=90) | Arm B: Dexamethasone + Melphalan (N=26) | Arm B: Dexamethasone + Cyclophosphamide (N=10) | Arm B: Dexamethasone + Thalidomide (N=1) | Arm B: Dexamethasone + Lenalidomide (N=47)
Abdominal distension (Gastrointestinal disorders) | 10 | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 9 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 7 | 4 | 2 | 0 | 9
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 0 | 1 | 0 | 2
Asthenia (General disorders) | 8 | 2 | 0 | 0 | 6
Atrial fibrillation (Cardiac disorders) | 6 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 3 | 1 | 0 | 5
Blood creatinine increased (Investigations) | 5 | 1 | 0 | 0 | 6
Bronchitis (Infections and infestations) | 8 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 7 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 6 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 18 | 3 | 4 | 1 | 13
Contusion (Injury, poisoning and procedural complications) | 6 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 0 | 2 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 11 | 3 | 2 | 0 | 4
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Depression (Psychiatric disorders) | 4 | 0 | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 32 | 4 | 1 | 0 | 22
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 14 | 3 | 1 | 0 | 7
Dizziness postural (Nervous system disorders) | 3 | 0 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 0 | 1 | 1
Dysaesthesia (Nervous system disorders) | 6 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 6 | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 7 | 1 | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 3 | 0 | 1 | 12
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 1 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 40 | 7 | 3 | 1 | 24
Flatulence (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 10 | 1 | 0 | 0 | 3
Herpes zoster (Infections and infestations) | 8 | 1 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 4
Hypertension (Vascular disorders) | 11 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0 | 1 | 0 | 2
Hypotension (Vascular disorders) | 3 | 1 | 1 | 0 | 4
Influenza (Infections and infestations) | 7 | 1 | 1 | 1 | 3
Influenza like illness (General disorders) | 8 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 32 | 3 | 2 | 1 | 8
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 5 | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3
Lacrimation increased (Eye disorders) | 5 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 6 | 1 | 0 | 0 | 4
Malaise (General disorders) | 2 | 1 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 5 | 0 | 0 | 0 | 2
Mood swings (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 | 1 | 0 | 1 | 7
Muscular weakness (Musculoskeletal and connective tissue disorders) | 12 | 1 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0 | 0 | 4
Myopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 1 | 4 | 0 | 3
Nausea (Gastrointestinal disorders) | 23 | 4 | 3 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 2
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 41 | 7 | 3 | 0 | 17
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 3
Orthostatic hypotension (Vascular disorders) | 6 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 5 | 1 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 7 | 0 | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 0 | 0 | 1 | 10
Peripheral swelling (General disorders) | 5 | 0 | 1 | 0 | 2
Platelet count decreased (Investigations) | 4 | 2 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 1 | 2 | 0 | 4
Pyrexia (General disorders) | 7 | 0 | 0 | 0 | 7
Rash macular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 | 1 | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 0 | 0 | 3
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 2 | 1 | 0 | 3
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 22 | 3 | 1 | 0 | 10
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 3 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 3
Vision blurred (Eye disorders) | 5 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 13 | 3 | 2 | 0 | 6
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 4
Weight increased (Investigations) | 6 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT01659658/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT01659658/SAP_001.pdf